CLINICAL TRIAL: NCT02871115
Title: Pilot Study of a Pharmacy Intervention for Older Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ryan Nipp, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-230
Record Dates: First submitted 2016-08-13; First posted 2016-08-18 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer; Lung Cancer; GI Cancer
Keywords: Cancer Care
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacy Intervention (Experimental): Patients randomized to the pharmacy intervention (PRIME) will undergo evaluation with a clinical pharmacist at their second or third chemotherapy infusion who will
  * Perform detailed medication reconciliation
  * Obtain allergy and vaccination history
  * Evaluate and document polypharmacy (number of medications)
  * Document their findings in the medical record and discuss their recommendations (in-person, phone call, email) with each patient's oncology team
  Interventions: Other: Pharmacy Intervention
- Usual Care (Active Comparator): Participants receiving Usual Oncology Care will not meet with the pharmacist unless indicated as part of their routine clinical care
  * Study staff will obtain all patient-reported measures from the patient.
  * Remind participant to complete self-report measures
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Pharmacy Intervention — Patients randomized to the pharmacy intervention (PRIME) will undergo evaluation with a clinical pharmacist at their second or third chemotherapy infusion who will: (1) perform detailed medication reconciliation and obtain allergy and vaccination history; (2) evaluate and document polypharmacy, potentially inappropriate medications, lack of appropriate medications; and (3) document their findings in the medical record and discuss their recommendations the oncology team.
  Arms: Pharmacy Intervention
Other: Usual Care — Participants receiving usual oncology care will not meet with the pharmacist unless indicated as part of their routine clinical care. Study staff will obtain all patient-reported measures from the patient.
  Arms: Usual Care

SUMMARY:
The purpose of this research study is to address the challenge of medication management for older patients undergoing treatment for cancer. The sponsor of this protocol is the Massachusetts General Hospital Cancer Center who is providing funding for this research study.

DETAILED DESCRIPTION:
The goals of the proposed study are: (1) to demonstrate the feasibility and acceptability of delivering PRIME (Pharmacist Reconciliation to Improve Medication Management in the Elderly) to older patients with breast, gastrointestinal, and lung cancers; and (2) to estimate the effect size (i.e. the magnitude of the difference between groups) of PRIME for improving medication management (e.g. accurate medication list, less polypharmacy, fewer potentially inappropriate medications) and achieving up-to-date vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Diagnosed with any stage breast, GI or lung cancer
* Panning to receive first-line chemotherapy at MGH
* Verbal fluency in English

Exclusion Criteria:

* Unwilling or unable to participate in the study
* Significant psychiatric, cognitive or other comorbid disease which the treating clinician believes prohibits informed consent or participation in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01-02 (Actual); Study Completion 2018-04-14 (Actual)

PRIMARY OUTCOMES:
Rates of study enrollment | 2 years
  To determine rates of study enrollment, we will assess the proportion of eligible patients who enroll in the study.

SECONDARY OUTCOMES:
Rates of Study Completion | 2 years
  To determine study completion rates, we will evaluate the proportion of patients enrolled who complete the study.
Rates of study satisfaction | 2 years
  To determine rates of study satisfaction, we will examine the proportion of participants who report satisfaction with the structure, timing and content of the study, using Likert-type scale responses.
Rates of Medication List Accuracy | Baseline to 4 weeks
  Compare rates of medication list accuracy (defined as concordance between the medical record and the medication list the patient reports taking) between study arms at 4 weeks following enrollment.
Change In The Number Of Medications | Baseline to 4 weeks
  Compare change in the number of medications (defined as the number of medications a patient is prescribed) between study arms from baseline to 4 weeks following enrollment.
Number Of Medications | Baseline to 4 weeks
  Compare the number of medications (defined as the number of medications a patient is prescribed) between study arms at 4 weeks following enrollment.
Rates of Polypharmacy | Baseline to 4 weeks
  Compare rates of polypharmacy (defined as five or more medications) 4 weeks following enrollment between study arms.
Change In The Number Of Potentially Inappropriate Medications | Baseline to 4 weeks
  Compare change in the number of potentially inappropriate medications between study arms from baseline to 4 weeks following enrollment.
Number Of Potentially Inappropriate Medications | Baseline to 4 weeks
  Compare the number of potentially inappropriate medications between study arms at 4 weeks following enrollment.
Rates Of Appropriate Pneumococcal Vaccinations | Baseline to 4 weeks
  Compare rates of appropriate pneumococcal vaccinations (as defined by the 2016 National Comprehensive Cancer Network [NCCN] guidelines) between study arms at 4 weeks.
Rates Of Appropriate Pneumococcal Vaccinations | Baseline to 8 weeks
  Compare rates of appropriate pneumococcal vaccinations (as defined by the 2016 National Comprehensive Cancer Network [NCCN] guidelines) between study arms at 8 weeks.
Rates Of Appropriate Influenza Vaccinations | Baseline to 4 weeks
  Compare rates of appropriate influenza vaccinations (as defined by the 2016 National Comprehensive Cancer Network [NCCN] guidelines) between study arms at 4 weeks.
Rates Of Appropriate Influenza Vaccinations | Baseline to 8 weeks
  Compare rates of appropriate influenza vaccinations (as defined by the 2016 National Comprehensive Cancer Network [NCCN] guidelines) between study arms at 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No